CLINICAL TRIAL: NCT03999502
Title: A Pilot Study to Evaluate the Feasibility and the Safety of an Endoluminal-suturing Device (Endoimna) as a Treatment of GERD.
Brief Title: Endomina Suturing Device as a Treatment of GERD.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2018/260
Record Dates: First submitted 2019-01-07; First posted 2019-06-26 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: GERD
Keywords: Endoscopy; Mini invasive
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The procedure will be performed under general anesthesia with tracheal intubation. Endomina will be introduced into the stomach over a guidewire and then fixed to the endoscope. The procedure will include at least one suture of the gastric cardia to tighten it. Patients will be kept overnight after the procedure.
  Interventions: Device: Endomina

INTERVENTIONS:
Device: Endomina — The procedure will be performed under general anesthesia with tracheal intubation. Endomina will be introduced into the stomach over a guidewire and then fixed to the endoscope. The procedure will include at least one suture of the gastric cardia to tighten it. Patients will be kept overnight after the procedure.

SUMMARY:
Gastroesophageal Reflux Disease (GERD) is a common problem affecting 10-20% of the population in the Western World.

Surgical therapy is able to restore the EGJ barrier function against reflux of the gastric content, decreases symptoms and improves the quality of life in GERD patients. However, there remain concerns regarding postoperative adverse events and the durability of the surgical procedure.

The ability to perform endoscopic full-thickness plications with Endomina-v2 will be used to assess safety and feasibility of the procedure in reducing GERD in patients suffering with chronic GERD, unsatisfied with PPIs, and/or complaining of persistent GERD symptoms despite PPI use.

DETAILED DESCRIPTION:
Gastroesophageal Reflux Disease (GERD) is a common problem affecting 10-20% of the population in the Western World. Approximately 250 million subjects worldwide and 30 million subjects in the US suffer from GERD. Among the 12 million Americans who suffer from daily heart-burn (the main symptom of GERD) almost 5 million do not respond completely to medications and many more do not want or cannot take medications due to side-effects (1). The goals of treatment in GERD are to relieve symptoms, heal esophagitis if present, prevent recurrence of symptoms and esophagitis, and prevent complications. Medical acid-suppressive therapy with proton pump inhibitors (PPIs) heals esophagitis, relieves symptoms and improves quality of life. However, acid suppressive therapy does not correct the underlying pathophysiology of dysfunction of the lower esophageal sphincter and hence symptoms of reflux due to weakly acidic or non-acid reflux persist in the majority of subjects who present with symptoms persisting on PPIs (regurgitations) (2).

Abnormalities in the structure and function of the esophago-gastric junction (EGJ) such as a permanently open EGJ, a hiatal hernia, a hypotensive lower esophageal sphincter (LES), and transient LES relaxations (t-LESR) are the main pathophysiologic mechanisms leading to GERD (3).

Surgical therapy is able to restore the EGJ barrier function against reflux of the gastric content, decreases symptoms and improves the quality of life in GERD patients (4,5). However, there remain concerns regarding postoperative adverse events and the durability of the surgical procedure (6,7). The results reported from operations performed in community hospital lower volume centers have been different than those achieved in centers of excellence. It has been reported that between 23% and 62% of patients who have undergone laparoscopic Nissen fundoplication use acid suppression medications at long-term follow-up. Due to these issues patient and physician acceptance of surgical procedures remains low and is mainly limited to patients with severe GERD or those non-responsive to medications. For these reasons, less invasive endoscopic techniques to treat GERD have been developed during the last 2 decades, which may be categorized into 3 groups: (1) sewing/plication at the cardia and EGJ, (2) radiofrequency (RF) thermal therapy to the LES, and (3) injection/implantation of biopolymers at the EGJ. Minimally invasive endoluminal procedures for GERD are designed to provide long-lasting symptom relief and abolish or lessen medication dependency. Most endoluminal modalities that were introduced into clinical practice have failed due to lack of long-term efficacy, complications, or interruption of commercialization due to financial difficulties of the companies that developed the techniques (8,9). Endoscopic sewing/plication techniques comprised mucosal plications (Endocinch) that were not clinically useful because the plications were not durable, and full-thickness (serosa-to-serosa) plications allowing prolonged durability (NDO Plicator device and Esophyx device). The data from the RCTs with Plicator device were encouraging and the finding of better results with multiple plications without an increase in adverse events supported that this device could have clinical utility. However, the company ceased operations in 2008 and the device is no longer clinically available (10). Transoral incisionless fundoplication (TIF) using Esophyx showed promising results in open studies (11). However, long-term follow-up revealed that a majority of patients required either ongoing PPI use or were referred for LNF owing to persistent symptoms (12).

Endomina-v2 (Endo Tools Therapeutics SA, Rue Auguste Piccard 48, 6041 GOSSELIES, Belgium) is a CE marked device that can be attached to an endoscope inside the body and allows manipulation of angulated tools during a peroral intervention. It offers the possibility to perform transoral surgical full thickness sutures and transoral endoscopic gastroplasty has shown to be safe and effective at mid-term follow-up in obese patients (13). The ability to perform endoscopic full-thickness plications with Endomina-v2 will be used to assess safety and feasibility of the procedure in reducing GERD in patients suffering with chronic GERD, unsatisfied with PPIs, and/or complaining of persistent GERD symptoms despite PPI use.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject is 21 - 70 years of age at the time of informed consent 2. Subject has documented symptoms of GERD (heartburn and/or regurgitation) for longer than 12 months, which respond at least partially to proton pump inhibitors (PPIs) 3. Subject is under continuous PPI therapy for at least 6 months 4. Subject has a diagnosis of GERD based on at least 2 of the following criteria:

  1. Past demonstration of reflux esophagitis grade A, B or C (LA classification)
  2. Abnormal esophageal acid exposure during esophageal pH-impedance monitoring (defined as distal esophageal pH < 4 for > 4 % of the monitoring time) performed after at least 7 days off of PPIs
  3. Positive symptom association between GERD symptoms and reflux episodes (symptom association probability ≥ 95%) demonstrated at pH-impedance monitoring)

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria cannot be enrolled in the study:

  1. Subject underwent previous surgery involving the gastroesophageal junction, such as a Nissen fundoplication
  2. Subject underwent previous endoscopic intervention for the treatment of GERD and/or Barrett's esophagus
  3. Subject has a hiatal hernia larger than 3 cm as determined by endoscopy
  4. Subject has history of gastroparesis
  5. Subject has any non-GERD esophageal motility disorders that in the opinion of investigator precludes an anti-reflux procedure
  6. Subject has history of or known esophageal stricture or significant esophageal anatomic abnormalities (obstructive lesions, etc.)
  7. Subject has Barrett's epithelium or any grade of dysplasia
  8. Subject has documented history of esophagitis Grade D (LA Classification)
  9. Subject has a history of suspected or confirmed esophageal or gastric cancer
  10. Subject has esophageal or gastric varices
  11. Subject has symptoms of dysphagia more than once per week every week within the last 3 months
  12. Subject is unable to tolerate withdrawal from PPI medications
  13. Subject has a body mass index (BMI) > 35 kg/m2
  14. Subject has any significant multisystem diseases
  15. Subject has an autoimmune or a connective tissue disorder (scleroderma, dematomyositis, Calcinosis-Raynaud's-Esophagus Sclerodactyly Syndrome (CREST), Sjogren's Syndrome, Sharp's Syndrome, etc.) requiring therapy in the preceding 2 years
  16. Subject has Type 1 diabetes mellitus or uncontrolled Type 2 diabetes mellitus (T2DM) defined as HbA1c > 9.5 in the previous 6 months or at screening/baseline
  17. Subject has had a significant cerebrovascular event within the last 6 months
  18. Female subject of child-bearing potential and is pregnant or nursing, or intends to become pregnant during the trial period, who is not using a reliable form of birth control
  19. Subject is currently enrolled in other potentially confounding research
  20. Subject has an active infection as determined by the investigator
  21. Subject has a history of any malignancy in the last 2 years
  22. Subject has a life expectancy less than 3 years
  23. Subject has a diagnosed major psychiatric disorder (bipolar, schizophrenia, etc.)
  24. Subject has any condition that, at the discretion of the investigator or sponsor, would interfere with accurate interpretation of the study endpoints or preclude participation in the trial
  25. Subject has a diagnosis of eosinophilic esophagitis

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-05-15 (Actual); Primary Completion 2021-05-12 (Estimated); Study Completion 2022-05-12 (Estimated)

PRIMARY OUTCOMES:
number of sutures at endoscopy (feasibility) | 12 months follow-up
  persistence of sutures at endoscopy
Incidence of all Adverse Device Effects | 12 months follow-up
  Safety will be characterized by the incidence of all Adverse Device Effects

SECONDARY OUTCOMES:
Assessment of Reflux (1) | 6 month follow-up
  Change from baseline to the 6-month follow-up visit of the mean percentage (%) of time distal esophageal pH is <4.0 using Esophageal Impedance-pH Monitoring performed of at least 7 days off PPIs and at least 2 days off H2 blocker
Assessment of Reflux (2) | 6 month follow-up
  Change from baseline to the 6-month follow-up visit of the total number of reflux episodes, proximal reflux episodes and DeMeester score using Esophageal Impedance-pH Monitoring
Evaluation of Esogastric junction | 6 month follow-up
  Change from baseline to the 6-month follow-up visit of the basal LES pressure and IRP4s using High resolution esophageal manometry
Gastro-esophageal reflux disease health-related quality of life score (GERD-HRQL score) | Baseline 3, 6 and 12 month follow-up
  Change from baseline to the 3, 6 and 12 months follow-up visit of the mean GERD-HRQL score. GERD-HRQL score has 13 items, which focus on heartburn symptoms, dysphagia, regurgitations, medication effects and the patient's present health condition. Each item is scored from 0 to 5, with a lower score indicating a better quality of life.
Reflux Symptom Index Score | Baseline 3, 6 and 12 month follow-up
  Change from baseline to the 3, 6 and 12 months follow-up visit of the mean Reflux Symptom Index (RSI) score. Reflux Symptom Index Score is an 9-item index designed to assess laryngo-pharyngeal symptoms related to gastro-esophageal reflux. Scores range from 0 to 5, with a higher score indicating more severe symptoms.
Mean acid-suppression medication use | Baseline 3, 6 and 12 month follow-up
  Mean acid-suppression (PPI and H2 blocker) medication use at 3, 6 and 12 months follow up.
Mean quality of life change | Baseline, 6 and 12 month follow-up
  Change from baseline to the 6 and 12 months follow-up visit of the Mean Quality of life scores as measured by SF-12. Twelve-Item Short-Form Health Survey (SF-12) is a multipurpose short form survey with 12 questions measuring physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality (energy/fatigue), social functioning, role limitations due to emotional problems, and mental health (psychological distress and well being). Norm-based scoring (NBS) linearly transforms the scales and summary measures to have a mean of 50 and standard deviation of 10 based on US general population data, so that a higher score indicates a better health state.

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology Department Erasme Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No